CLINICAL TRIAL: NCT01977742
Title: A Sudden Rest-exercise Transition Training to Improve Cardiac Vagal Tone
Brief Title: Rest-exercise Transition Training to Improve Cardiac Vagal Tone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Medicina do Exercício (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 191.2011-15/12/11
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Subjects Evaluated With Low Cardiac Vagal Tone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initiate with SEP but without RTTE (Active Comparator): Initiate supervised exercise (SEP) program but without rest-exercise transition training (RTTE)to improve cardiac vagal tone at same time; will stop RTTE after 8 weeks.
  Interventions: Other: Supervised exercise program; Other: Supervised exercise program together with a specific sudden rest-exercise training protocol
- Initiate with RETT and SEP (Active Comparator): Supervised exercise program (aerobic, strength and flexibility exercises) and a specific sudden rest-exercise training protocol, three times a week. After 8 weeks, the sudden rest-exercise training protocol will be discontinued.
  The cardiac vagal index will be measured at every 8 weeks.
  Interventions: Other: Supervised exercise program; Other: Supervised exercise program together with a specific sudden rest-exercise training protocol

INTERVENTIONS:
Other: Supervised exercise program — Aerobic, strength and flexibility exercises in a supervised exercise program for 8 weeks; after 8 weeks will add a specific sudden rest-exercise training protocol, three times a week. The cardiac vagal index will be measured at every 8 weeks.
Other: Supervised exercise program together with a specific sudden rest-exercise training protocol — Aerobic, strength and flexibility exercises in a supervised exercise program for 8 weeks together with a specific sudden rest-exercise training protocol, three times a week After 8 weeks will discontinue the specific sudden rest-exercise training protocol. The cardiac vagal index will be measured at every 8 weeks.

SUMMARY:
Purpose: to investigate the hypothetical additive value of a sudden rest-exercise training over the cardiac vagal of cardiac patients in a supervised exercise program.

DETAILED DESCRIPTION:
Allocating in the admission for a supervised exercise program all subjects evaluated with low cardiac vagal tone (cardiac vagal index ≤ 1,30), it is expected that from a sample of almost 150 subjects (all over 18 years-old, ranging mostly from 40 to 50), we will compare 50 subjects that adhered to the supervised exercise program ( more than 65% of expected presence). Patients with pacemaker on unable to exercise in the bicycle will be excluded from the study, as well as those who does not adhere to at least more than 65% of the expected presence in the supervised exercise program.

All the sample will be randomized to performed 8 weeks of a specific sudden rest-exercise training and after 8 weeks will discontinue the protocol, or will do the opposite ( 8 weeks of no specific protocol, followed by 8 weeks of specific sudden rest-exercise training). The cardiac vagal will be evaluated at every 8 weeks to measure the cardiac vagal index between both phases. During all the time, all clients will perform aerobic, strength and flexibility exercises as part of the supervised exercise program.

ELIGIBILITY:
Inclusion Criteria:

* cardiac vagal index ≤ 1,30

Exclusion Criteria:

* pacemaker
* low adherence
* cognitive/physical impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Supervised exercise program and rest-exercise transition training to improve cardiac vagal tone | 16 weeks
  Cardiac vagal tone after either 8 weeks of aerobic, strength and flexibility exercises alone or 8 weeks of aerobic, strength, flexibility exercises combined with specific sudden rest-exercise training

SECONDARY OUTCOMES:
Longitudinal effects of supervised exercise program and rest-exercise transition training to improve cardiac vagal tone | 1 year
  Cardiac vagal tone measures at every 8 weeks after both phases (16 weeks of training / no training, depending of the randomization) during a year

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gil S Araujo, PhD, Principal Investigator — Gama Filho University